CLINICAL TRIAL: NCT07318792
Title: Evaluation of the Safety and the Clinical Effectiveness of Using Tropocells® Autologous PRF System to Treat Chronic, Non-healing, Non-infected Wounds in Combination With Standard of Care (SOC).
Brief Title: Using TropoCells(R) Autologous Platelet-Rich Fibrin (PRF) to Treat Chronic Non-Healing Wounds
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Estar Medical dba Medical Technologies, LTD (Industry)
Collaborators: Global Clinical Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RND054- AIM II Chronic Wounds
Record Dates: First submitted 2026-01-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Wound Chronic Draining; Wound Closure
Keywords: Chronic Non-healing Wounds; TropoCells(R) Platelet-rich Fibrin (PRF); Autologous Platelet-rich Fibrin (PRF); Platelet Derived Therapy

STUDY DESIGN:
Intervention Model Description: Non-randomized, Single group
Masking Description: No parties are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participants with non-infected, mild-to-moderate, chronic open soft tissue wound (Active Comparator): Tropocells® Autologous Platelet-Rich Fibrin (PRF) to be topically applied for the management of exuding cutaneous wounds, such as leg ulcers, pressure ulcers, and diabetic ulcers and mechanically or surgically debrided wounds", intended to be used at point-of-care for the safe and rapid preparation of platelet-rich plasma (PRP) gel from a small sample of a patient's own peripheral blood. Under the supervision of a healthcare professional.
  Interventions: Device: Platelet-rich fibrin (PRF)

INTERVENTIONS:
Device: Platelet-rich fibrin (PRF) — Standard of Care will include-
  1. Nutritional Supplementation using 14 days Juven(R)
  2. Wound Cleansing and Debridement
  3. Mild to Moderate Compression as needed for edema Control
  4. Off-loading as needed (foot gear, chair cushions, bed mattresses)
  5. Antimicrobial Dressings as needed
  6. Edema Control
  7. Negative Pressure Wound Therapy- as needed
  8. Collagen dressings as indicated
  9. Optimized perfusion/oxygenation
  10. Treated Underlying Medical Conditions

SUMMARY:
Platelet-based therapies have been used to treat bony and soft tissue effects for more than 30 years. Tropocells® Autologous Platelet-Rich Fibrin (PRF) is being used to treat chronic, non-healing wounds, of a variety of types. This will help determine the safety and effective use of PRF in the treatment of soft tissue defects.

DETAILED DESCRIPTION:
Chronic wounds are wounds that fail to progress through a normal healing process in a timely fashion. Typically the wounds remain in a pro-inflammatory state. The activation of platelets reacting to tissue damage initiates most healing sequences. The use of activated platelets in the form or platelet-rich plasma (PRP) and/or platelet-rich fibrin (PRF) applied to a clean wound base has been associated with improved wound healing outcomes for bony and soft tissues, especially when associated with standard of care (SOC), including supporting underlying medical conditions, improved perfusion and oxygenation, edema control, removing recurrent insults for trauma, treating infection, and preventing ongoing inflammatory triggers. Activated platelets in the form of Tropocells(R) autologous platelet-rich fibrin (PRF) made from "blood drawn from peripheral veins, and centrifuged into a gel, topically applied to exuding cutaneous wounds such as leg ulcers, pressure ulcers and diabetic ulcers, and mechanically or surgically-debrided wounds." Sixteen (16) Subjects will be enrolled to evaluate the efficacy and safety when used to treat chronic noninfected, nonhealing, mild to moderately ischemic wounds.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ≥ 18≤ 80 years of age 2. Chronic wounds present for at least thirty (30) days meeting classification as, mild to moderate severity, open exuding wound, including, leg ulcer, pressure ulcer, or mechanically or surgically debrided.

  3. Located in any anatomical location on the body. 4. If more than one non-healing wound is present, an index wound will be selected ≥ 1.0 cm2 size and less than or equal to 25.0 cm2.

  5. If the wound is in an ulcer cluster the dominant ulcer will be selected, with at least 2.0 cm2 between the index wound and other wounds.

  6. The study wound will be present for at least thirty (30) days and the subject will have undergone standard of care assessment and intervention, according to the wound type being evaluated, where SOC may include, but not be limited to, proper cleansing and debridement, off-loading, compression, bioburden reduction, moisture management, infection control, optimized perfusion, venous ablation, nutrition supplementation, smoking cessation counseling and medical therapy, and access to wound and underlying disease education and training.

  7. Neurovascular assessment, conducted according to the assessment typically performed for the wound type will be performed during Screening (Study Visit 1), and repeated at the level normally conducted at the follow-up visits. Perfusion should be adequate to sustain a healing process. Neurological examinations will be performed to document the presence of neuropathy and/or nerve injury.

  8. Documented 40% or less wound closure during thirty (30) days of standard of care (SOC).

  9. No clinical signs of infection at the wound site or the affected limb. 10. Post-debridement with no residual necrotic tissue. 11. Platelet counts should be within normal range ≥ 105,000 to <450, 000. 12. Hemoglobin (Hgb) ≥ 10 g/dL and Hematocrit (HCT) ≥ 27%. 13. HbA1C ≤ 12%. 14. Chronic renal failure (CRF) and dialysis patients may be enrolled. 15. PT/aPTT/INR should be within normal limits unless the subject is on coumadin, then maintain range of INR 2 to 3.

  16. Prealbumin ≥ 15 mg/dL. 17. Adequate off-loading of the wound site for wheelchair bound, bed bound, and ambulatory subjects.

  18. Multi-layered compression dressings for venous related wounds. 19. Females of childbearing potential should not be pregnant and agree to avoid conceiving during the study.

  20. Males agree to use contraception or abstinence during the study. 21. The subject has provided written informed consent prior to any screening procedures and agrees to comply with study procedures and requirements.

  22. Usual care therapies that may be included will be negative pressure wound therapy (NPWT), antimicrobial dressings, collagen containing matrix and packing materials.

Exclusion Criteria:

* Exclusion Criteria

  1. Life expectancy is less than twelve (12) months.
  2. Participation in another clinical trial involving an investigational device or drug within thirty (30) days prior to enrollment.
  3. Sepsis within two (2) weeks prior to enrollment.
  4. Soft tissue infection affecting the wound within two (2) weeks prior to enrollment.
  5. Known osteomyelitis or occult osteomyelitis documented with inﬂammatory markers ESR ≥ 60 and/or CRP ≥7.9 mg/dL.
  6. Religious constraints to using blood products, including autologous blood.
  7. Alcohol or substance abuse (other than tobacco) within 2 months prior.
  8. Severe lymphedema at Stage 3b or greater (lymphostatic elephantiasis).
  9. The inability to use compression therapy for venous insufficiency or lymphedema.
  10. Subjects who are cognitively impaired, unable to understand the informed consent, or have a health care proxy.
  11. Hemophilia, sickle cell anemia, thrombocytopenia, and leukemia or blood dyscrasia.
  12. History of problems with coagulation, abnormal thrombocytes (platelets), or receiving heparin, intravenously. However, subjects taking coumadin, aspirin, clopidogrel, or other oral anti-coagulants are not excluded.
  13. Cytostatic therapy within the past 12 months.
  14. The subject has inadequate venous access for repeated blood draw.
  15. Known HBV, HCV, or HIV.
  16. Blood-borne or communicable disease that would likely prevent full participation in the trial (HIV, AIDS, COVID-19).
  17. Subjects with known sensitivity to blood components of the PRF Kit (e.g., rubber stopper, vacutainer tubing).
  18. Advanced therapy treatments with hyperbaric oxygen, electrical stimulation (eStim), pulsed electromagnetic energy fields (PEMF), colored light therapies, cellular tissue products (CTPs) like amniotic tissues, Apligraf® and Dermagraft® will be excluded; while NPWT, collagen matrix products (sheet or bulk packing), antimicrobial dressings (surfactants, silver or copper, hypochlorous acid) may be used.

AIDS- acquired immunodeficiency syndrome; COPD-chronic obstructive pulmonary disease; COVID-19- Coronavirus Disease-19; CRP- C-reactive protein; ESR-erythrocyte sedimentation rate; HBV-hepatitis B virus; HCV- hepatitis C virus; HIV- human immune-deficiency virus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | From Screening to end of follow-up at 9 weeks
  Number of Subjects with Complete Wound Closure- defined as 100% re-epithelialization remaining closed during two (2) consecutive weekly follow-up assessments.
  * Intent-to-treat analysis
  * Per-protocol analysis

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MCR Health-Advanced Specialty Institute (ASI), Bradenton, Florida
  - San Antonio Vascular and Endovascular Clinic (SAVE), San Antonio, Texas
  - The San Antonio Vascular and Endovascular Clinic (SAVE), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data will be shared with the FDA in support of the IDE, if required. There is no plan to share IPD with journals or publications.

REFERENCES:
- [Background] Bolton L. Platelet-Rich Plasma: Optimal Use in Surgical Wounds. Wounds. 2021 Aug;33(8):219-221. PMID 34357880
- [Background] Milek T, Nagraba L, Mitek T, Wozniak W, Mlosek K, Olszewski W, Ciostek P, Deszczynski J, Kuchar E, Stolarczyk A. Autologous Platelet-Rich Plasma Reduces Healing Time of Chronic Venous Leg Ulcers: A Prospective Observational Study. Adv Exp Med Biol. 2019;1176:109-117. doi: 10.1007/5584_2019_388. PMID 31134552
- [Background] Qu W, Wang Z, Hunt C, Morrow AS, Urtecho M, Amin M, Shah S, Hasan B, Abd-Rabu R, Ashmore Z, Kubrova E, Prokop LJ, Murad MH. The Effectiveness and Safety of Platelet-Rich Plasma for Chronic Wounds: A Systematic Review and Meta-analysis. Mayo Clin Proc. 2021 Sep;96(9):2407-2417. doi: 10.1016/j.mayocp.2021.01.030. Epub 2021 Jul 3. PMID 34226023
- [Background] Meznerics FA, Fehervari P, Dembrovszky F, Kovacs KD, Kemeny LV, Csupor D, Hegyi P, Banvolgyi A. Platelet-Rich Plasma in Chronic Wound Management: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. J Clin Med. 2022 Dec 19;11(24):7532. doi: 10.3390/jcm11247532. PMID 36556151
- [Background] 1. Wounds International: White paper on wound balance - Achieving wound healing with confidence (2023), https://woundsinternational.com/wp-content/uploads/2023/04/HAR23_Supp_Wound-Balance_WINT-Web.pdf.